CLINICAL TRIAL: NCT03121911
Title: Effects of Interval Physical Training on Inflammatory Markers, Cardiac Autonomic Modulation at Rest, Expiratory Flow Limitation and Respiratory Efficiency in Recent Myocardial Infarction
Brief Title: Effects of Interval Physical Training on Expiratory Flow Limitation in Recent Myocardial Infarction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: technical problems in equipment
Sponsor: Federal University of Uberlandia (Other)
Collaborators: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Débora Lara Zuza Scheucher, Principal Investigator, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 005040/2017
Record Dates: First submitted 2017-04-06; First posted 2017-04-20 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Expiratory Flow Limitation; Recent Myocardial Infarction
Keywords: Recent Myocardial Infarction; Interval Physical Training; Inspiratory Muscle Training; Expiratory Flow Limitation; Ventilatory Efficiency; Inflammatory Markers; Heart Rate Variability
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: 54 patients will be included, divided into three groups with 18 participants each. All will be submitted to several exams applied to the monitoring of cardiac and pulmonary function. Then, groups 1 (IT) and group 2 (IT + IMT) will participate in a physical training program for 12 weeks and will be re-evaluated after this period. In addition, they will be monitored for a 6 month period after discharge, with returns every two months to measure the energy expenditure through an accelerometer, and at the end of this period they will repeat all the tests again. Group 3 (absence of CR), will consist of patients who do not live in the city or those who can not participate in the CR program for any other reason, and will only participate in the evaluations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - Interval Training (IT) (Experimental): All participants will be submitted to several exams of cardiac and pulmonary functions. Then, group 1 (IT) will participate in a physical training program for 12 weeks and will be re-evaluated after this period. After discharge, they will be monitored for an aditional period of 6 months, with returns every two months to measure the energy expenditure (accelerometer). At the end of this period all the tests will be repeated.
  Each exercise session will last for 60 minutes and will be divided into three parts as follows: warm up (10 minutes); interval training (IT) - 30 minutes of IT performed in a cycle ergometer, divided into 6 levels of intensity based on the ventilatory anaerobic threshold found in CPET (70%, 80%, 100% and 110%); cooling down (10 minutes).
  Interventions: Other: Interval Training (IT)
- Group 2 - IT + IMT (Experimental): All participants will be submitted to the same evaluations before and after training, and 6 months after discharge. Group 2 (IT + inspiratory muscle training (IMT)) will participate in a 12 week physical training program. After discharge, they will be monitored for an aditional period of 6 months, with returns every two months to measure the energy expenditure.
  The group 2 will perform the IMT session at the end of the warm-up exercises, prior to the beginning of the IT on a cycloergometer. IMT session consists of 2 series of 12 inspirations with a 60% of MIP. Participant will be asked to inhale quickly and deeply, as quickly as possible, with a 2 minutes interval between series. All the others exercises will be identical between group 1 and 2.
  Interventions: Other: Interval Training (IT); Other: Inspiratory Muscle Training (IMT)
- Group 3 - Absence of rehabilitation (No Intervention): Group 3 (absence of rehabilitation) will be made up of those patients who for any reason do not agree to participate in the rehabilitation program, such as those who do not live in the city, and will remain without intervention. All participants in this group will perform all the evaluations procedures, comprised of: heart rate variability, hematological and biochemical profile, erythrocytes membrane deformability and stability, inflammatory markers, respiratory pressures, plethysmography, spirometry, carbon monoxide diffusion capacity, ankle brachial index, electrical bioimpedance, echocardiogram, quality of life questionnaires (SF-36 and MacNew QLMI), cardiopulmonary exercise testing and constant load tests.

INTERVENTIONS:
Other: Interval Training (IT) — Each exercise session will consist of:
  1. warm up (10 minutes)- stretches and calisthenics exercises of low to moderate intensity;
  2. interval training (IT) - 30 minutes of IT performed in a cycle ergometer, divided into 6 levels of intensity based on the ventilatory anaerobic threshold (VAT) found in CPET: Level 1 - 5 minutes in moderate intensity, at 80% of power reached in VAT; Levels 2 and 4 - 5 minutes of moderate to high intensity, at 100% of VAT; Levels 3 and 5 - 5 minutes of moderate to high intensity, 110% of VAT; Level 6 - 5 minutes in moderate intensity, at 70% of VAT.
  3. cooling down (10 minutes) - stretching, and breathing exercises. An CPET will be performed every four weeks to adjust the intensity of training.
  Arms: Group 1 - Interval Training (IT); Group 2 - IT + IMT
Other: Inspiratory Muscle Training (IMT) — The IMT session will take place just after the warm-up exercises and consist of 2 series of 12 inspirations with a 60% of Maximal Inspiratory Pressure (MIP) with the equipment POWERbreathe Plus Medic® (POWERbreathe International Ltd, Warwickshire, UK). The patient will be instructed to remain seated with a nasal clip during the IMT series to avoid nasal air leakage and will be asked to inhale quickly and deeply, as quickly as possible, with a 2 minute interval between series. The training load will be adjusted weekly by a new evaluation of MIP to maintain the intensity of the exercise within the proposed value.
  All the others exercises will be identical between group 1 and 2.
  Arms: Group 2 - IT + IMT

SUMMARY:
Introduction: Expiratory flow limitation (EFL) and ventilatory inefficiency during dynamic exercise have been identified in patients with recent myocardial infarction (RMI) with preserved ventricular and pulmonary function. However, it is not known what is the prevalence of EFL in this population and what are the effects of physical and respiratory training on this limitation.

Objectives: To evaluate the prevalence of EFL and ventilatory inefficiency during dynamic exercise in individuals with uncomplicated RMI, and to evaluate the effects of interval physical training (IT) in addition to inspiratory muscle training (IMT), exclusive IT and absence of cardiopulmonary rehabilitation (CR) on EFL and ventilatory efficiency.

Methods: 54 patients will be included, divided into three groups with 18 participants each. All will be submitted to evaluations of heart rate variability, hematological and biochemical profile, erythrocytes membrane deformability and stability, inflammatory markers, respiratory pressures, plethysmography, spirometry, carbon monoxide diffusion capacity, ankle brachial index, electrical bioimpedance, echocardiogram, quality of life questionnaires, cardiopulmonary exercise testing and constant load tests. Then, groups 1 (IT) and group 2 (IT + IMT) will participate in a physical training program for 12 weeks and will be re-evaluated after this period. In addition, they will be monitored for a 6 month period after discharge, with returns every two months to measure the energy expenditure through an accelerometer, and at the end of this period they will repeat all the tests again. Group 3 (absence of CR), will consist of patients who do not live in the city or those who can not participate in the CR program for any other reason, and will only participate in the evaluations.

DETAILED DESCRIPTION:
Patients with coronary artery disease (CAD) attended by the Sistema Unico de Saude (SUS) in the city of Uberlandia and region are routinely referred to Hospital de Clinicas - Federal University of Uberlandia after acute myocardial infarction (AMI) for coronary angiography and other exams, receiving appropriate clinical or surgical follow-up. After the resolution of the clinical condition, the patient is released from the hospital with a medical referral to the Cardiorespiratory Rehabilitation Program offered by the institution.

These patients are contacted by telephone by the team of the rehabilitation sector, and invited to attend for a pre-entry evaluation for inclusion in treatment. In this telephone contact the secretary of the sector clarifies that the hospital does not have transportation services for the patients who accept to be part of the program, and afterwards the evaluation is scheduled. The initial anamnesis will be performed by a multidisciplinary team. In this screening are collected complaints, past and current history of possible diseases, personal and family history, life habits, medications in use, exams performed pre-hospital discharge and physical examination, collected from an individual anamnesis form. At the end of the evaluation the patient receives a card with the scheduling of training days that occur three times a week and dressing and feeding instructions prior to training.

All volunteers who fit the study criteria will be invited to participate in the study, being informed about the experimental procedures to which they would be submitted. They will also be clarified that all the information collected during the accomplishment of the work will be kept confidential, protecting their identities. Individuals who agree to participate in the study will sign an informed consent according to National Health Council (466/12) guidelines, and a next return will be scheduled to begin physical testing and blood collection. At that moment, the Research Participant Identification Card will be filled in, which will be kept in a confidential place separated from the other evaluations, with restricted access to the researcher, and a code will be given to the participant. In case of refusal to participate in the study, the participant will receive the same care offered to other patients routinely referred to the rehabilitation sector, being included into the conventional rehabilitation program that also lasts for 12 weeks.

Considering that the patients enrolled in the research will have to attend for evaluation and monitoring related to the study, all the displacements related to these additional activities will be refunded to the participants during the entire period of the study.

The evaluation procedures that will be performed in 2 days will consist of: Step 1 - ankle brachial index, heart rate variability at rest, respiratory pressures (maximal inspiratory and expiratory pressures), cardiopulmonary exercise test (incremental and constant load tests), spirometry and quality of life questionnaires (SF-36 and MacNew QLMI); Step 2 - blood collection (hematological and biochemical profile, erythrocytes membrane deformability and stability, inflammatory markers), plethysmography, carbon monoxide diffusion capacity and echocardiography.

After these exams the participant will be randomized to a training group: Group 1 - interval training (IT) or group 2 - IT + inspiratory muscle training (IMT), and will participate in the cardiorespiratory rehabilitation program for a period of 12 weeks, three times a week. Group 3 will consist of those participants who for any reason do not agree to participate in the rehabilitation program, such as those who do not live in the city, and will remain without intervention.

During the 6 months of discharge, participants will be monitored monthly, by telephone contact to verify possible changes in medications in use and general health status.

At the end of the 2nd, 4th and 6th month of discharge, in the last week of each period, the patient will be invited to return to the rehabilitation sector for placement of an accelerometer, a monitor that quantifies free activities and sedentary lifestyle. The selected equipment (activPAL3 ™ micro, PAL Technologies Ltd, Scotland, UK) makes use of algorithms properties to quantify periods of sitting, orthostatism and walking. This information will be used to estimate the daily energy expenditure in the period and will store information of seven consecutive days during the selected weeks.

The re-evaluations will consist of all the exams mentioned above (steps 1 and 2), and will be performed at the beginning and at the end of the training period and after 6 months of the program's discharge.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Aged 35 to 80 years
* Recent myocardial infarction (RMI), between 15 and 45 days post-event, being the 1st MI event
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Preserved respiratory muscle strength (Maximal Inspiratory Pressure > 60% predicted)
* Whether or not submitted to Percutaneous Transluminal Coronary Angioplasty (PTCA)
* Presence of expiratory flow limitation by incremental cardiopulmonary test
* Agreement to participate in the study after reading and signing the informed consent

Non-inclusion Criteria:

* Body Mass Index (BMI) ≥ 35 kg / m2
* Previous diagnosis of any musculoskeletal, neurological, respiratory or vascular diseases
* Ankle Brachial Index (ABI) < 0.90 and > 1.4
* Diabetes mellitus
* Active or smoking cessation for less than six months
* Chronic organic dysfunction such as renal or hepatic impairment
* Patients submitted to Coronary Artery Bypass Graft Surgery (CABG)
* Inadequate response of systemic or electrocardiographic blood pressure during the cardiopulmonary exercise test (CPET)
* Presence of Chronic Obstructive Pulmonary Disease (COPD) or Interstitial Lung Diseases
* Presence of valvulopathies or Chagas disease
* Participants with pacemaker (PM) or implantable cardioverter defibrillator (ICD)

Exclusion Criteria:

* Refusal to participate in the study
* Participants who do not complete all the steps proposed in the research
* Participants who request their exclusion at any time during the study, will be excluded

Ages: 35 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Change on Expiratory Flow Limitation (EFL) | Change from baseline EFL, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation program
  Two constant workload exercise tests (CWET) will evaluate the EFL and the ventilatory strategy at the VAT and VAT + 25%, with rest interval of 30 to 60 minutes between tests.
  Duration: 20 minutes each test. Patients will be monitored with optoelectronic plethysmography and transthoracic electrical cardioimpedance. After a 2-minute rest period in a cycle ergometer (clinical evaluation, metabolic, cardiovascular, ventilatory and gas exchange records, and Borg), the effort will start at zero load (60 rpm). The pre-established intensity corresponding to VAT and 25% above VAT will be placed in the 3rd minute of exercise by single increment for ten minutes. In the last four minutes the flow-volume loops will be measured. After each test there will be an active recovery for 3 minutes, and 2 minutes of rest.
  EFL will be evaluated by comparing tidal flow-volume loops, obtained after an inspiratory capacity maneuver, with the resting maximal flow-volume loop measured before each CWET.

SECONDARY OUTCOMES:
Change on Ankle Brachial Index (ABI) | Change from baseline ABI, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation program
  To this exam will be used a Doppler ultrasound (Portable Vascular Doppler; DV610B; MEDMEGA, Brazil), gel and sphygmomanometer.
  Volunteers will be instructed to remain at rest in the supine position for ten minutes. The cuff will be positioned 3 cm above the cubital fossa in the upper limbs and 3 cm above the medial malleolus in the lower limbs, considering the correct alignment to the arterial path. A 45 to 60º angle will be observed between the skin and the Doppler transducer in the opposite direction to the blood flow in order to amplify the sound of the signal. Systolic arterial pressures will be measured in the 4 limbs: right brachial artery; right posterior tibial and dorsalis pedis arteries; left posterior tibial and dorsalis pedis arteries; and left brachial artery.
  The ABI will be calculated as the ratio between the highest of the two systolic pressures below the ankle (posterior tibial and dorsalis pedis artery) with the highest brachial portion pressure.
Change on Heart Rate Variability (HRV) at rest | Change from baseline HRV, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation program
  This test will evaluate the autonomic modulation of the heart rate response from its variability (HRV) during rest in the supine, orthostatic and sitting positions. For this, the volunteers will be monitored with a cardiofrequencymeter (Polar Electro ™, V800 ™, OY, Kempele, Finland) and thoracic belt.
  Participants will be instructed to remain at rest, with a normal quiet breathing and not to talk during the examination. After 600 seconds of supine rest, HR will be collected for another 600 seconds in each position: supine, standing and sitting positions.
  Data recorded will be transferred to a computer via FlowSync ™ software. The data will be inspected visually, and for each volunteer, the sequence of RR interval (ms) with 256 consecutive beats will be selected at the time of greater signal stability. Subsequently, the linear and non-linear analysis of the HRV will be performed.
Change on Maximal Inspiratory Pressure (MIP) | Change from baseline MIP, once a week during the training period, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation program
  A digital manovacuometer (MVD300®, Globalmed, Porto Alegre, RS, Brazil) will be used to perform the respiratory pressures, with an operating range of ± 300 cmH2O.
  The volunteer will be seated with feet resting on the floor, and will receive instruction on how to proceed during the test. A nasal clip will be positioned five seconds before performing the maneuver to avoid air leaks, and the patient will be asked to press the cheeks with the hands. The volunteer will be instructed to close the lips firmly around the buccal, to exhale all the air until reaching the residual volume (RV) and to make a forced inspiration for approximately one to two seconds. Each patient will perform three maneuvers with 2-minute rest intervals between the replicates. If the last maneuver is greater than the previous ones, a further measurement will be made. The highest value will be used for the analyzes. Static values lower than 60% of predicted will be considered as respiratory muscle weakness.
Change on Maximal Expiratory Pressure (MEP) | Change from baseline MEP, once a week during the training period, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation program
  The equipment for performing MEP will be the same as described for MIP, as well as patient positioning. The PE max will be measured from the total lung capacity (TLC), using a nasal clip, and the volunteer will be asked for a maximal expiratory effort sustained for one to two seconds. At least three maneuvers with 2-minute rest intervals between the replicates will be performed, using the highest value for the analyzes. If the last maneuver is greater than the previous ones, a further measurement will be made, and so on until the last value is not greater than the previous one. MEP minimum value of normality for men is 150 cmH2O.
Change on Incremental Cardiopulmonary Exercise Testing (CPET) | Change from baseline CPET, every 4 weeks during the training period, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation
  Objective: evaluate the aerobic power; identify the VAT and the HR response. Variables measured respiration by respiration, will be: oxygen consumption, carbon dioxide production, respiration exchange ratio, minute ventilation, respiratory rate, ventilatory equivalent (O2 and CO2), end-tidal tensions of oxygen and carbon dioxide, inspiratory and expiratory time and total time of respiratory cycle.
  Duration: 8 - 12 minutes. After a 2-minute rest period (clinical evaluation, metabolic, cardiovascular, ventilatory and gas exchange records, and Borg evaluation), the effort will start at zero load (60 rpm) and increase at the 2nd minute of exercise until the maximum tolerance. Exhaustion will be noticed as malaise, lipothymia, nausea, extreme dyspnea (Borg 10) or chest pain expressed by the patient. The test will also be ended in the presence of fatigue (< 60 rpm) or maximum HR. After interruption of the increment, will start a 3-minute period of zero load and 2 minutes of rest.
Change on Spirometry | Change from baseline spirometry, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation
  Before and after each constant workload exercise tests (CWET), spirometry will be performed using the Clinical Pulmonary Function-Spirometry (CPF-S™, Medical Graphics Corporation, St. Paul, MN- USA). Pre-CWET spirometry will be used to identify the reference variables at rest for the maximal flow-volume loop (MFVL) to allow comparison with the values during CWET. Post-CWET spirometry has the purpose to evaluate the presence of exercise-induced bronchodilation.
Change on Medical Outcome Study 36-item Short Form Health Survey (SF-36) | Change from baseline SF-36, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation
  In the rest interval between the CWET, the quality of life questionnaires will be administered in the interview format.
  The generic SF-36 will be used in order to quantify the function and general well-being of the patient, allowing the comparison between different populations and studies.
  The questionnaire consists of the physical and mental components, encompassing a total of eight domains: physical component that involves (1) functional capacity (question 3), (2) pain (questions 7 and 8), (3) general health status (1 and 11) and (4) physical aspect (question 4); And mental component that includes (5) mental health (9B, C, D, F, H), (6) emotional aspect (question 5), (7) social aspect (questions 6 and 10) and (8) vitality (9A, E, G, I). Each domain has a final score of 0 to 100, with zero worse health status and 100, better health status.
Change on MacNew Heart Disease Health-related Quality of Life Questionnaire (MacNew QLMI) | Change from baseline MacNew QLMI, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation
  In the rest interval between the CWET, the quality of life questionnaires will be administered in the interview format.
  The MacNew specific questionnaire will reveal functional symptoms and limitations attributed to the myocardial infaction, being more sensitive to changes in the clinical condition as results from the interventions. It consists of 27 items that fall into three domains: physical limitation (13 items), emotional function (14 items) and social function (13 items).
Change on Bioelectrical Impedance Analysis (BIA) | Change from baseline BIA, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation
  BIA aims to assess body composition by quantifying water in tissues. Before beginning the procedure, volunteers will be instructed to empty the urinary bladder and remove any metallic objects in contact to the body. They will then be placed in rest in the supine position for 10 minutes, with abduction of upper and lower limbs, forming an angle of at least 30 ° to avoid any contact between the limbs. The distal electrode will be placed in the right hand and right foot. The two distal electrodes (black clips) will be placed on the dorsal surface of the hand (metacarpophalangeal of the middle finger) and the foot (metatarsophalangeal of the middle finger), while current collectors (proximal red clips) will be applied in the styloid process, above the joint line of the wrist and between the medial and lateral malleoli of the ankle, above the joint interline.
  These proximal electrodes collect the voltage drop due to impedance, assigning values to the body composition.
Change on Blood collection - hematological parameters | Change from baseline Blood Collection, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation
  After a 12 hour fasting, the blood will be collected by venipuncture in evacuated tubes (Vacuntainer®) containing specific anticoagulants, and analyzed by the Clinical Analysis Laboratory of the Clinical Hospital - Federal University of Uberlandia (FUU). Hematological parameters: complete blood count, lipid profile, glucose, folic acid, CRP, glycated hemoglobin, vitamin B12, serum iron, ferritin, transferrin capacity index, uric acid, albumin, lactate dehydrogenase, reticulocytes, total, direct and indirect bilirubin.
Change on Blood collection - erythrocyte membrane stability | Change from baseline Blood Collection, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation
  After a 12 hour fasting, the blood will be collected by venipuncture in evacuated tubes (Vacuntainer®) containing specific anticoagulants.
  To erythrocyte membrane stability, a sample with EDTA will be sent to the Laboratory of Biophysiochemistry (FUU), and another to the Laboratory of Biochemistry (FUU) for analysis of oxidative stress.
Change on Blood collection - inflammatory markers | Change from baseline Blood Collection, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation
  After a 12 hour fasting, the blood will be collected by venipuncture in evacuated tubes (Vacuntainer®) containing specific anticoagulants, and analyzed by the Clinical Analysis Laboratory of the Clinical Hospital - Federal University of Uberlandia (FUU).
  A sample without anticoagulant will be sent to the Laboratory of Nanobiotechnology (FUU) for analysis of inflammatory markers and another to the Laboratory Eduardo Mineiro for homocysteine analysis. The required amount of blood for all the analyzes shall be 31 ml.
Change on Plethysmography parameters - residual capacity (FRC) | Change from baseline plethysmography, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation
  Static pulmonary volume measurements will be performed using the full-body plethysmography Elite Platinum DX system (Medical Graphics Corporation, St. Paul, MN, USA). The patient, within the hermetically sealed plethysmographic enclosure, will be instructed to make small, uniform, repetitive breathing movements against an obstruction at the airway opening at a frequency of 60 Hz. This maneuver aims to establish the starting point in functional residual capacity (FRC).
Change on Plethysmography parameters - residual volume (RV) | Change from baseline plethysmography, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation
  The gas in the lungs is alternately compressed and decompressed, and such changes in thoracic volume are reflected by inverse variations of the thoracic cage, which is reflected by changes in pressure in the interior of the plethysmographic cabin.
  Indirectly, the residual volume (RV) is calculated using a vital capacity (VC) maneuver done immediately afterwards to estimate the lung capacity of each patient.
Change on Plethysmography parameters - total pulmonary capacity (TPC) | Change from baseline plethysmography, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation
  The gas in the lungs is alternately compressed and decompressed, and such changes in thoracic volume are reflected by inverse variations of the thoracic cage, which is reflected by changes in pressure in the interior of the plethysmographic cabin.
  Indirectly, the total pulmonary capacity (TPC) is calculated using a vital capacity (VC) maneuver done immediately afterwards to estimate the lung capacity of each patient.
Change on Carbon Monoxide Diffusion Capacity (DLCO) | Change from baseline DLCO, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation
  DLCO analyzes the amount of carbon monoxide (CO) that diffuses to the pulmonary capillaries through the alveolar-capillary barrier. The system used for this evaluation will be Elite Platinum DX (Medical Graphics Corporation-MGC, MN, USA), applying the modified Krogh technique (single breathing).
  The patient will inhale a test gas (0.3% CO, 10% Helium, 21% O2 balanced with nitrogen) and will sustain in the lungs a volume corresponding to 90% of the VC for 10 seconds. During expiration, tracer gas (Helium) concentrations, with an inert (no diffusion) characteristic, and CO, will be continuously analyzed by a rapid response analyzer. Thus, the amount of exhaled CO is measured by determining the amount to be diluted in the lungs (estimated by tracer gas concentration), and thus the difference in relation to the inhaled concentration (previously known) indicates the total that will diffuse by the alveolar-capillary membrane.
Change on Echocardiography (ECHO) | Change from baseline ECHO, after 12 weeks at the end of the rehabilitation program and 6 months after release from rehabilitation
  Echocardiogram performed during hospitalization will be used as an inclusion criteria (LVEF ≥ 50%). The purpose of the exam will be to monitor the evolution of left ventricular function in response to the implemented therapies and to correlate it with the other tests performed. All ECHO will be performed in the Echocardiography Sector (FUU), by a properly trained professional of the institution.
Accelerometer - Energy expenditure | At the end of the 2nd, 4th and 6th month of discharge from the rehabilitation program, in the last week of each period.
  At the end of the 2nd, 4th and 6th month of discharge from the rehabilitation program, in the last week of each period, the patient will be invited to return for placement of an accelerometer, a monitor that quantifies free activities and sedentary lifestyle. The selected equipment (activPAL3™ micro, PAL Technologies Ltd, Scotland, UK) makes use of algorithm properties to quantify periods of sitting, standing and walking. This information will be used to estimate the daily energy expenditure in the period and will store information for seven consecutive days during the selected weeks.
  The microactivPAL3™ will be packed in a nitrile glove and attached to the skin by tegaderm™ (3M, Sumaré, SP) so that the patient can bathe with the device. The data will be transmitted to the computer via USB input (activPAL3 ™ micro USB port docking station, PAL Technologies Ltd, Scotland, UK) and analyzed by activPAL ™ software (PAL Technologies Ltd, Scotland, UK).

CONTACTS AND LOCATIONS:
Overall Officials: Debora LZ Scheucher, M.S., Principal Investigator — Federal University of Uberlandia
Locations (1):
- Universidade Federal de Uberlândia, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Angadi SS, Mookadam F, Lee CD, Tucker WJ, Haykowsky MJ, Gaesser GA. High-intensity interval training vs. moderate-intensity continuous exercise training in heart failure with preserved ejection fraction: a pilot study. J Appl Physiol (1985). 2015 Sep 15;119(6):753-8. doi: 10.1152/japplphysiol.00518.2014. Epub 2014 Sep 4. PMID 25190739
- [Background] Antila K. Quantitative characterization of heart rate during exercise. Scand J Clin Lab Invest Suppl. 1979;(153):3-68. No abstract available. PMID 293886
- [Background] Arend M, Kivastik J, Maestu J. Maximal inspiratory pressure is influenced by intensity of the warm-up protocol. Respir Physiol Neurobiol. 2016 Aug;230:11-5. doi: 10.1016/j.resp.2016.05.002. Epub 2016 May 12. PMID 27181328
- [Background] Arnold SV, Spertus JA, Jones PG, Xiao L, Cohen DJ. The impact of dyspnea on health-related quality of life in patients with coronary artery disease: results from the PREMIER registry. Am Heart J. 2009 Jun;157(6):1042-9.e1. doi: 10.1016/j.ahj.2009.03.021. PMID 19464415
- [Background] Aulin J, Siegbahn A, Hijazi Z, Ezekowitz MD, Andersson U, Connolly SJ, Huber K, Reilly PA, Wallentin L, Oldgren J. Interleukin-6 and C-reactive protein and risk for death and cardiovascular events in patients with atrial fibrillation. Am Heart J. 2015 Dec;170(6):1151-60. doi: 10.1016/j.ahj.2015.09.018. Epub 2015 Oct 3. PMID 26678637
- [Background] Billat LV. Interval training for performance: a scientific and empirical practice. Special recommendations for middle- and long-distance running. Part I: aerobic interval training. Sports Med. 2001;31(1):13-31. doi: 10.2165/00007256-200131010-00002. PMID 11219499
- [Background] Baba R, Nagashima M, Goto M, Nagano Y, Yokota M, Tauchi N, Nishibata K. Oxygen uptake efficiency slope: a new index of cardiorespiratory functional reserve derived from the relation between oxygen uptake and minute ventilation during incremental exercise. J Am Coll Cardiol. 1996 Nov 15;28(6):1567-72. doi: 10.1016/s0735-1097(96)00412-3. PMID 8917273
- [Background] Balady GJ, Arena R, Sietsema K, Myers J, Coke L, Fletcher GF, Forman D, Franklin B, Guazzi M, Gulati M, Keteyian SJ, Lavie CJ, Macko R, Mancini D, Milani RV; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Interdisciplinary Council on Quality of Care and Outcomes Research. Clinician's Guide to cardiopulmonary exercise testing in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 13;122(2):191-225. doi: 10.1161/CIR.0b013e3181e52e69. Epub 2010 Jun 28. No abstract available. PMID 20585013
- [Background] Barbosa-Silva MC, Barros AJ, Wang J, Heymsfield SB, Pierson RN Jr. Bioelectrical impedance analysis: population reference values for phase angle by age and sex. Am J Clin Nutr. 2005 Jul;82(1):49-52. doi: 10.1093/ajcn.82.1.49. PMID 16002799
- [Background] Black LF, Hyatt RE. Maximal respiratory pressures: normal values and relationship to age and sex. Am Rev Respir Dis. 1969 May;99(5):696-702. doi: 10.1164/arrd.1969.99.5.696. No abstract available. PMID 5772056
- [Background] Caruso P, Albuquerque AL, Santana PV, Cardenas LZ, Ferreira JG, Prina E, Trevizan PF, Pereira MC, Iamonti V, Pletsch R, Macchione MC, Carvalho CR. Diagnostic methods to assess inspiratory and expiratory muscle strength. J Bras Pneumol. 2015 Mar-Apr;41(2):110-23. doi: 10.1590/S1806-37132015000004474. PMID 25972965
- [Background] Conraads VM, Pattyn N, De Maeyer C, Beckers PJ, Coeckelberghs E, Cornelissen VA, Denollet J, Frederix G, Goetschalckx K, Hoymans VY, Possemiers N, Schepers D, Shivalkar B, Voigt JU, Van Craenenbroeck EM, Vanhees L. Aerobic interval training and continuous training equally improve aerobic exercise capacity in patients with coronary artery disease: the SAINTEX-CAD study. Int J Cardiol. 2015 Jan 20;179:203-10. doi: 10.1016/j.ijcard.2014.10.155. Epub 2014 Oct 25. PMID 25464446
- [Background] Cornish AK, Broadbent S, Cheema BS. Interval training for patients with coronary artery disease: a systematic review. Eur J Appl Physiol. 2011 Apr;111(4):579-89. doi: 10.1007/s00421-010-1682-5. Epub 2010 Oct 23. PMID 20972578
- [Background] Masterson Creber RM, Lee CS, Margulies K, Riegel B. Identifying biomarker patterns and predictors of inflammation and myocardial stress. J Card Fail. 2015 Jun;21(6):439-45. doi: 10.1016/j.cardfail.2015.02.006. Epub 2015 Feb 26. PMID 25727486
- [Background] Fang L, Moore XL, Dart AM, Wang LM. Systemic inflammatory response following acute myocardial infarction. J Geriatr Cardiol. 2015 May;12(3):305-12. doi: 10.11909/j.issn.1671-5411.2015.03.020. PMID 26089856
- [Background] Ankle Brachial Index Collaboration; Fowkes FG, Murray GD, Butcher I, Heald CL, Lee RJ, Chambless LE, Folsom AR, Hirsch AT, Dramaix M, deBacker G, Wautrecht JC, Kornitzer M, Newman AB, Cushman M, Sutton-Tyrrell K, Fowkes FG, Lee AJ, Price JF, d'Agostino RB, Murabito JM, Norman PE, Jamrozik K, Curb JD, Masaki KH, Rodriguez BL, Dekker JM, Bouter LM, Heine RJ, Nijpels G, Stehouwer CD, Ferrucci L, McDermott MM, Stoffers HE, Hooi JD, Knottnerus JA, Ogren M, Hedblad B, Witteman JC, Breteler MM, Hunink MG, Hofman A, Criqui MH, Langer RD, Fronek A, Hiatt WR, Hamman R, Resnick HE, Guralnik J, McDermott MM. Ankle brachial index combined with Framingham Risk Score to predict cardiovascular events and mortality: a meta-analysis. JAMA. 2008 Jul 9;300(2):197-208. doi: 10.1001/jama.300.2.197. PMID 18612117
- [Background] Guazzi M, Arena R, Guazzi MD. Evolving changes in lung interstitial fluid content after acute myocardial infarction: mechanisms and pathophysiological correlates. Am J Physiol Heart Circ Physiol. 2008 Mar;294(3):H1357-64. doi: 10.1152/ajpheart.00866.2007. Epub 2008 Jan 11. PMID 18192218
- [Background] Guzzetti S, Borroni E, Garbelli PE, Ceriani E, Della Bella P, Montano N, Cogliati C, Somers VK, Malliani A, Porta A. Symbolic dynamics of heart rate variability: a probe to investigate cardiac autonomic modulation. Circulation. 2005 Jul 26;112(4):465-70. doi: 10.1161/CIRCULATIONAHA.104.518449. Epub 2005 Jul 18. PMID 16027252
- [Background] Haensel A, Mills PJ, Nelesen RA, Ziegler MG, Dimsdale JE. The relationship between heart rate variability and inflammatory markers in cardiovascular diseases. Psychoneuroendocrinology. 2008 Nov;33(10):1305-12. doi: 10.1016/j.psyneuen.2008.08.007. Epub 2008 Sep 25. PMID 18819754
- [Background] Ho KK, Moody GB, Peng CK, Mietus JE, Larson MG, Levy D, Goldberger AL. Predicting survival in heart failure case and control subjects by use of fully automated methods for deriving nonlinear and conventional indices of heart rate dynamics. Circulation. 1997 Aug 5;96(3):842-8. doi: 10.1161/01.cir.96.3.842. PMID 9264491
- [Background] Huikuri HV, Makikallio TH, Perkiomaki J. Measurement of heart rate variability by methods based on nonlinear dynamics. J Electrocardiol. 2003;36 Suppl:95-9. doi: 10.1016/j.jelectrocard.2003.09.021. PMID 14716599
- [Background] Karsten M, Neves LM, Neves VR, Beltrame T, Borghi-Silva A, Arena R, Agostoni P, Catai AM. Recent myocardial infarction patients present ventilatory limitation during aerobic exercise. Int J Cardiol. 2012 Nov 29;161(3):180-1. doi: 10.1016/j.ijcard.2012.06.026. Epub 2012 Jun 22. No abstract available. PMID 22727969
- [Background] Nakajima KM, Rodrigues RC, Gallani MC, Alexandre NM, Oldridge N. Psychometric properties of MacNew Heart Disease Health-related Quality of Life Questionnaire: Brazilian version. J Adv Nurs. 2009 May;65(5):1084-94. doi: 10.1111/j.1365-2648.2009.04962.x. Epub 2009 Mar 9. PMID 19291183
- [Background] Neder JA, Andreoni S, Lerario MC, Nery LE. Reference values for lung function tests. II. Maximal respiratory pressures and voluntary ventilation. Braz J Med Biol Res. 1999 Jun;32(6):719-27. doi: 10.1590/s0100-879x1999000600007. PMID 10412550
- [Background] Neder JA, Andreoni S, Peres C, Nery LE. Reference values for lung function tests. III. Carbon monoxide diffusing capacity (transfer factor). Braz J Med Biol Res. 1999 Jun;32(6):729-37. doi: 10.1590/s0100-879x1999000600008. PMID 10412551
- [Background] Neves LM, Karsten M, Neves VR, Beltrame T, Borghi-Silva A, Catai AM. Relationship between inspiratory muscle capacity and peak exercise tolerance in patients post-myocardial infarction. Heart Lung. 2012 Mar-Apr;41(2):137-45. doi: 10.1016/j.hrtlng.2011.07.010. Epub 2011 Dec 15. PMID 22177761
- [Background] Neves LM, Karsten M, Neves VR, Beltrame T, Borghi-Silva A, Catai AM. Respiratory muscle endurance is limited by lower ventilatory efficiency in post-myocardial infarction patients. Braz J Phys Ther. 2014 Jan-Feb;18(1):1-8. doi: 10.1590/s1413-35552012005000134. Epub 2014 Feb 1. PMID 24675907
- [Background] Oldridge N. Exercise-based cardiac rehabilitation in patients with coronary heart disease: meta-analysis outcomes revisited. Future Cardiol. 2012 Sep;8(5):729-51. doi: 10.2217/fca.12.34. PMID 23013125
- [Background] Palmefors H, DuttaRoy S, Rundqvist B, Borjesson M. The effect of physical activity or exercise on key biomarkers in atherosclerosis--a systematic review. Atherosclerosis. 2014 Jul;235(1):150-61. doi: 10.1016/j.atherosclerosis.2014.04.026. Epub 2014 May 1. PMID 24835434
- [Background] Pinkstaff S, Peberdy MA, Kontos MC, Fabiato A, Finucane S, Arena R. Usefulness of decrease in oxygen uptake efficiency slope to identify myocardial perfusion defects in men undergoing myocardial ischemic evaluation. Am J Cardiol. 2010 Dec 1;106(11):1534-9. doi: 10.1016/j.amjcard.2010.07.034. Epub 2010 Oct 14. PMID 21094351
- [Background] Porta A, Guzzetti S, Montano N, Furlan R, Pagani M, Malliani A, Cerutti S. Entropy, entropy rate, and pattern classification as tools to typify complexity in short heart period variability series. IEEE Trans Biomed Eng. 2001 Nov;48(11):1282-91. doi: 10.1109/10.959324. PMID 11686627
- [Background] Porta A, Tobaldini E, Guzzetti S, Furlan R, Montano N, Gnecchi-Ruscone T. Assessment of cardiac autonomic modulation during graded head-up tilt by symbolic analysis of heart rate variability. Am J Physiol Heart Circ Physiol. 2007 Jul;293(1):H702-8. doi: 10.1152/ajpheart.00006.2007. Epub 2007 Feb 16. PMID 17308016
- [Background] Prado DM, Rocco EA, Silva AG, Silva PF, Lazzari JM, Assumpcao GL, Thies SB, Suzaki CY, Puig RS, Furlan V. The influence of aerobic fitness status on ventilatory efficiency in patients with coronary artery disease. Clinics (Sao Paulo). 2015 Jan;70(1):46-51. doi: 10.6061/clinics/2015(01)09. PMID 25672429
- [Background] Prado DM, Rocco EA, Silva AG, Rocco DF, Pacheco MT, Furlan V. Effect of exercise training on ventilatory efficiency in patients with heart disease: a review. Braz J Med Biol Res. 2016 Jun 20;49(7):e5180. doi: 10.1590/1414-431X20165180. PMID 27332771
- [Background] 2011 WRITING GROUP MEMBERS; 2005 WRITING COMMITTEE MEMBERS; ACCF/AHA TASK FORCE MEMBERS. 2011 ACCF/AHA Focused Update of the Guideline for the Management of patients with peripheral artery disease (Updating the 2005 Guideline): a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2011 Nov 1;124(18):2020-45. doi: 10.1161/CIR.0b013e31822e80c3. Epub 2011 Sep 29. No abstract available. PMID 21959305
- [Background] Shepherd CW, While AE. Cardiac rehabilitation and quality of life: a systematic review. Int J Nurs Stud. 2012 Jun;49(6):755-71. doi: 10.1016/j.ijnurstu.2011.11.019. Epub 2011 Dec 23. PMID 22197653
- [Background] Takahashi AC, Porta A, Melo RC, Quiterio RJ, da Silva E, Borghi-Silva A, Tobaldini E, Montano N, Catai AM. Aging reduces complexity of heart rate variability assessed by conditional entropy and symbolic analysis. Intern Emerg Med. 2012 Jun;7(3):229-35. doi: 10.1007/s11739-011-0512-z. Epub 2011 Jan 21. PMID 21253879
- [Background] Tamburus NY, Paula RF, Kunz VC, Cesar MC, Moreno MA, da Silva E. Interval training based on ventilatory anaerobic threshold increases cardiac vagal modulation and decreases high-sensitivity c-reative protein: randomized clinical trial in coronary artery disease. Braz J Phys Ther. 2015 Nov-Dec;19(6):441-50. doi: 10.1590/bjpt-rbf.2014.0124. Epub 2015 Oct 9. PMID 26647745
- [Background] Anderson L, Oldridge N, Thompson DR, Zwisler AD, Rees K, Martin N, Taylor RS. Exercise-Based Cardiac Rehabilitation for Coronary Heart Disease: Cochrane Systematic Review and Meta-Analysis. J Am Coll Cardiol. 2016 Jan 5;67(1):1-12. doi: 10.1016/j.jacc.2015.10.044. PMID 26764059
- [Background] Van de Veire NR, Van Laethem C, Philippe J, De Winter O, De Backer G, Vanderheyden M, De Sutter J. VE/VCO2 slope and oxygen uptake efficiency slope in patients with coronary artery disease and intermediate peakVO2. Eur J Cardiovasc Prev Rehabil. 2006 Dec;13(6):916-23. doi: 10.1097/01.hjr.0000238400.35094.72. PMID 17143123
- [Background] von Kanel R, Carney RM, Zhao S, Whooley MA. Heart rate variability and biomarkers of systemic inflammation in patients with stable coronary heart disease: findings from the Heart and Soul Study. Clin Res Cardiol. 2011 Mar;100(3):241-7. doi: 10.1007/s00392-010-0236-5. Epub 2010 Sep 21. PMID 20857123